CLINICAL TRIAL: NCT00440102
Title: Ketamine Versus Etomidate During Rapid Sequence Intubation: Consequences on Hospital Morbidity
Acronym: KETASED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P060213
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2007-05

CONDITIONS: Intubation; Difficult
Keywords: ETOMIDATE; KETAMINE; RAPID SEQUENCE INTUBATION; PREHOSPITAL; During rapid sequence intubation
MeSH Terms: interventions — Ketamine; Etomidate

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): ketamine
  Interventions: Drug: Ketamine
- 2 (Active Comparator): Etomidate
  Interventions: Drug: Etomidate

INTERVENTIONS:
Drug: Ketamine — Ketamine
  Arms: 1
Drug: Etomidate — Etomidate
  Arms: 2

SUMMARY:
The expected benefit is a reduction of the morbidity of patients admitted in the intensive care unit having received ketamine for intubation.

DETAILED DESCRIPTION:
The national recommendations of sedation concerning the intubation in emergency settings advise the use of a hypnotic, etomidate associated to succinylcholine. A national inquiry showed that more than 80% of prehospital intubations use a rapid sequence intubation as sedation. However, several recent studies throw into question the use of etomidate in this indication. Indeed, etomidate is a powerful inhibitor of the synthesis of cortisol. Adrenocortical hormone insufficiency is clearly associated to an increase in the morbidity-mortality of critically ill patients. Several authors advise therefore against the use of etomidate for such patients. Yet, to date, only indirect arguments associating the use of etomidate with excessive morbidity-mortality exist. A real causality link is not yet established. Another hypnotic that could constitute a therapeutic alternative to the use of etomidate exists: ketamine. The advantage of this molecule is that it does not inhibit the adrenocortical hormone axis.

Objectives: To evaluate sedation using ketamine versus etomidate in term of morbidity-mortality in critically ill patients intubated in the prehospital setting.

Experimental diagram: A prospective, multicentric, randomized, controlled, simple blind trial with independent analysis of the primary outcome.

The expected benefit is a reduction of the morbidity of patients admitted in the intensive care unit having received ketamine for intubation. The risks incurred for patients being suitable to this research are bound essentially to the adverse effects of ketamine. These include some psycho-dyslectic manifestations: nightmare, unpleasant awakening, and disruption of the visual, auditory sensations and mood, a sensation to float and sometimes depersonalization. These adverse effects are warned by a continuous administration of benzodiazepines.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring sedation for prehospital endotracheal intubation
* Age ≥ 18 years
* Consent of a family member if present, then of the patient for the pursuit of research

Exclusion Criteria:

* Patient in cardiac arrest
* Presence of contraindication to succinylcholine:

  * Personal or familial history of malignant hyperthermia
  * Known hypersensitivity to succinylcholine
  * Skeletal muscle disease
  * Myasthenia
  * Known hyperkalemia
  * Severe ophthalmic injury
  * Known congenital deficit in plasmatic pseudo-cholinesterase
* Presence of contraindication to ketamine:

  * Known hypersensitivity to ketamine
  * Known porphyria
  * Severe hypertension
* Presence of contraindication to etomidate:

  * Known untreated adrenal insufficiency
  * Known hypersensitivity to etomidate
* Known pregnancy
* Unaffiliated patient to the social insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Maximal value of the "Sepsis-related Organ Failure" Assessment (SOFA) | at the end of D2

SECONDARY OUTCOMES:
Mortality, length of stay in the intensive care unit and in the hospital, length of stay under artificial ventilation, neurological state at the exit of the hospital and adverse effects : within the first 28 days. | at D0
intubation difficulty | at D0
early complications | at D0
adverse effects | at D0
SOFA in the first 48 hours of hospitalization | at the ende of D2

CONTACTS AND LOCATIONS:
Overall Officials: Frederic ADNET, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Chu Avicenne, Bobigny, France

REFERENCES:
- [Result] Jabre P, Combes X, Lapostolle F, Dhaouadi M, Ricard-Hibon A, Vivien B, Bertrand L, Beltramini A, Gamand P, Albizzati S, Perdrizet D, Lebail G, Chollet-Xemard C, Maxime V, Brun-Buisson C, Lefrant JY, Bollaert PE, Megarbane B, Ricard JD, Anguel N, Vicaut E, Adnet F; KETASED Collaborative Study Group. Etomidate versus ketamine for rapid sequence intubation in acutely ill patients: a multicentre randomised controlled trial. Lancet. 2009 Jul 25;374(9686):293-300. doi: 10.1016/S0140-6736(09)60949-1. Epub 2009 Jul 1. PMID 19573904
- [Result] Wenzel V, Lindner KH. Best pharmacological practice in prehospital intubation. Lancet. 2009 Jul 25;374(9686):267-8. doi: 10.1016/S0140-6736(09)61071-0. Epub 2009 Jul 1. No abstract available. PMID 19573905